CLINICAL TRIAL: NCT05694871
Title: Official Title A Randomized Phase 2 Trial With a Safety Lead-In to Evaluate Palbociclib Versus Palbociclib and Cemiplimab for the Treatment of Advanced Dedifferentiated Liposarcoma
Brief Title: Testing the Addition of Cemiplimab to Palbociclib for the Treatment of Advanced Dedifferentiated Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A092107; NCI-2022-08568 (Other: NCI)
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Dedifferentiated Liposarcoma; Locally Advanced Dedifferentiated Liposarcoma; Metastatic Dedifferentiated Liposarcoma; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IV Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Unresectable Dedifferentiated Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — palbociclib; cemiplimab; Immunoglobulin G; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (palbociclib) (Active Comparator): Patients receive palbociclib PO on study. Patients will be allowed to cross over to Arm II following documentation of disease progression. Patients undergo MRI or CT scans throughout the trial. Patients may also undergo blood sample collection on study.
  Interventions: Drug: Palbociclib; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Procedure: Biospecimen collection; Other: Questionnaire Administration
- Arm II (palbociclib, cemiplimab) (Experimental): Patients receive palbociclib PO and cemiplimab IV on study. Patients undergo MRI or a CT scan throughout the trial. Patients may also undergo blood sample collection on study.
  Interventions: Drug: Palbociclib; Biological: Cemiplimab; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Procedure: Biospecimen collection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Palbociclib — Given PO
  Other Names: PD-0332991
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Immunoglobulin G4
  Arms: Arm II (palbociclib, cemiplimab)
Procedure: Magnetic Resonance Imaging — undergo MRI
  Other Names: MRI
Procedure: Computed Tomography — Undergo a CT Scan
  Other Names: CAT Scan; CT Scan
Procedure: Biospecimen collection — Undergo blood sample collection
Other: Questionnaire Administration — Ancillary Studies

SUMMARY:
This phase II trial compares the effect of treatment with palbociclib alone to treatment with palbociclib plus cemiplimab for treating patients with dedifferentiated liposarcoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Palbociclib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Cemiplimab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. The combination of these two drugs may be more effective in shrinking or stabilizing advanced dedifferentiated liposarcoma compared to palbociclib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform a safety lead-in among 6 patients to confirm that the combination of palbociclib and cemiplimab is safe and tolerable.

II. To evaluate whether palbociclib in combination with cemiplimab (Arm 2) demonstrates a superior progression-free survival (PFS) compared to palbociclib monotherapy (Arm 1) for patients with advanced dedifferentiated liposarcoma (DDLPS).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile in and across each treatment arm as determined by both Common Terminology Criteria for Adverse Events (CTCAE) and Patient Reported Outcomes (PRO)-CTCAE criteria.

II. To evaluate and compare the objective response rate (ORR) and duration of response (DOR) in and across each treatment arm.

III. To evaluate and compare the overall survival (OS) in and across each treatment arm.

IV. To evaluate and compare progression-free rate at 8 weeks (PFR8) in and across each treatment arm.

EXPLORATORY OBJECTIVES:

I. To collect genomic sequencing data previously collected as standard of care, including data on CDK4 copy number (as determined by fluorescence in situ hybridization [FISH] or other molecular testing).

II. To conduct multiplex immunohistochemistry using archival tumor tissue (where available) to define densities of infiltrating immune cell subsets and tumor and immune cell major histocompatibility complex (MHC) and PD-L1 expression.

III. To perform an exploratory analysis to evaluate for any relationship between CDK4 copy number and (a) the tumor immune microenvironment as defined by multiplex immunohistochemistry and (b) clinical outcomes from study treatment.

IV. To explore efficacy and toxicity endpoints, including PFS and ORR, for patients who progress on palbociclib monotherapy and crossover to the palbociclib plus cemiplimab combination.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive palbociclib orally (PO) on study. Patients will be allowed to cross over to Arm II following documentation of disease progression. Patients undergo magnetic resonance imaging (MRI) or computed tomography (CT) scans throughout the trial. Patients may also undergo blood sample collection on study.

ARM II: Patients receive palbociclib PO and cemiplimab intravenously (IV) on study. Patients undergo MRI or CT scans throughout the trial. Patients may also undergo blood sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA (STEP 1): Patients must have histologically documented dedifferentiated liposarcoma (DDLPS). Patients with mixed well-differentiated/dedifferentiated liposarcoma (WD/DD LPS) tumors are eligible provided there is a histologically confirmed DDLPS component at some point during the treatment course

  * Disease must be metastatic or locally advanced and surgically unresectable, in the opinion of the treating investigator
  * Note: Intact retinoblastoma protein (RB) can be assumed in DDLPS. In a query of project Genomics Evidence Neoplasia Information Exchange (GENIE) (American Association for Cancer Research [AACR]), including 286 DDLPS tumors, the rate of RB1 mutation in DDLPS was 1.37%. Therefore, molecular testing to determine intact Rb is not required
* ELIGIBILITY CRITERIA (STEP 1): Patients must have at least one lesion that is measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria to be eligible for this study. Previously radiated lesions should not be used as target lesions unless there is documented evidence of disease progression of that lesion after radiation
* ELIGIBILITY CRITERIA (STEP 1): Patients may have received any number of prior systemic treatment lines for DDLPS, including none
* ELIGIBILITY CRITERIA (STEP 1): Patients must have recovered to baseline or =< grade 1 per CTCAE version 5.0 from toxicity related to any prior treatment, unless adverse events are clinically nonsignificant and/or stable on supportive therapy, and with the exceptions of fatigue (which must be =< grade 2), alopecia and/or endocrinopathies related to prior immunotherapy which are controlled with hormone replacement
* ELIGIBILITY CRITERIA (STEP 1): Patients must have completed all prior anti-cancer treatment, including radiation, >= 14 days prior to registration
* ELIGIBILITY CRITERIA (STEP 1): Age >= 18 years
* ELIGIBILITY CRITERIA (STEP 1): Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* ELIGIBILITY CRITERIA (STEP 1): Absolute neutrophil count (ANC) >= 1000/mm^3
* ELIGIBILITY CRITERIA (STEP 1): Platelet count >= 100,000/mm^3
* ELIGIBILITY CRITERIA (STEP 1): Hemoglobin >= 9 g/dL
* ELIGIBILITY CRITERIA (STEP 1): Creatinine clearance (CrCl) >= 30 mL/min
* ELIGIBILITY CRITERIA (STEP 1): Total bilirubin =< 1.5 x upper limit of normal (ULN)
* ELIGIBILITY CRITERIA (STEP 1): Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x ULN
* ELIGIBILITY CRITERIA (STEP 1): Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible, patients should be class IIB or better. Furthermore, patients may not have an uncontrolled ventricular arrhythmia or recent (within 3 months) myocardial infarction
* ELIGIBILITY CRITERIA (STEP 1): For patients with evidence of chronic hepatitis B (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* ELIGIBILITY CRITERIA (STEP 1): Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently receiving treatment, they are eligible if they have an undetectable HCV viral load
* ELIGIBILITY CRITERIA (STEP 1): Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* ELIGIBILITY CRITERIA (STEP 1): Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Patients participating on this trial may not be receiving other anti-neoplastic therapies and there should be no anticipated need for such therapy
* ELIGIBILITY CRITERIA (STEP 1): Patients with treated brain metastases that are non-progressing are eligible if follow-up brain imaging performed at least 4 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are not eligible
* ELIGIBILITY CRITERIA (STEP 1): Patients must be able to swallow oral medications
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR STEP 2 CROSSOVER FROM ARM 1 TO ARM 2): In order to cross over to Arm 2, patients must meet the same eligibility criteria as described above
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR STEP 2 CROSSOVER FROM ARM 1 TO ARM 2): Patients must have demonstrated progression of disease on palbociclib monotherapy (Arm 1) per RECIST version 1.1 criteria

Exclusion Criteria:

* ELIGIBILITY CRITERIA (STEP 1): Patients may not have received prior treatment with CDK4/6 inhibitors (including, but not limited to: palbociclib, ribociclib or abemaciclib) or anti-PD-1/anti-PD-L1 antibodies
* ELIGIBILITY CRITERIA (STEP 1): Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects

  * Therefore, for women of childbearing potential only, a negative serum pregnancy test done =< 7 days prior to registration is required
* ELIGIBILITY CRITERIA (STEP 1): Patients must not have an active autoimmune disease with the exception of vitiligo, well-controlled asthma or allergic rhinitis, type 1 diabetes, psoriasis or hypothyroidism. Patients with a history of adrenal insufficiency are eligible if on a stable dose of prednisone =< 10 mg or equivalent
* ELIGIBILITY CRITERIA (STEP 1): Patients must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any other condition that would limit compliance with study requirements
* ELIGIBILITY CRITERIA (STEP 1): Patients may not require the use of chronic steroids in excess of 10 mg prednisone daily or equivalent
* ELIGIBILITY CRITERIA (STEP 1): Patients may not require concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir). The required washout period prior to re-registration 2 weeks
* ELIGIBILITY CRITERIA (STEP 1): Patients may not require concomitant use of known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort). The required washout period prior to re-registration is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR STEP 2 CROSSOVER FROM ARM 1 TO ARM 2): Patients may not have experienced a grade 3 or higher non-hematologic adverse event deemed clinically significant in the opinion of the treating investigator, or have discontinued palbociclib due to toxicity, while participating on Arm 1

  * Patients must also have recovered to baseline or =< grade 1 per CTCAE version 5.0 from toxicity related to Arm 1 treatment, unless adverse events are clinically nonsignificant and/or stable on supportive therapy, and with the exceptions of fatigue (which must be =< grade 2), alopecia and/or endocrinopathies related to prior immunotherapy which are controlled with hormone replacement
  * Note: Patients who underwent dose reduction of palbociclib during treatment on Arm 1 will begin treatment on Arm 2 at the same dose (i.e. dose re-escalation is not allowed)
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR STEP 2 CROSSOVER FROM ARM 1 TO ARM 2): Patients may not have received prior treatment with anti-PD-1/anti-PD-L1 antibodies
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR STEP 2 CROSSOVER FROM ARM 1 TO ARM 2): Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects * Therefore, for women of childbearing potential only, a negative serum pregnancy test done =< 7 days prior to re-registration is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The time from randomization to the first documentation of disease progression or death, assessed up to 48 months.
  Efficacy analyses will be based on intention to treat principles. PFS will be compared between the two treatment arms using Kaplan-Meier methods. The hazard ratio, median PFS, and estimated PFS rates at 12, 24, 36, and 48 months will be estimated along with corresponding 95% confidence intervals. A log-rank test will be used to compare the PFS distributions between the two treatment arms in this cohort. Cox proportional hazards models will also be used to assess the impact of treatment arm on PFS when stratifying on the stratification factors.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Patients will be evaluated for adverse events using the National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0. Summary statistics (e.g., mean, median, standard deviation) and frequency tables will be used to describe the distributions of adverse events. Rates of adverse events occurring in the treatment arm will be compared to the control arm with chi-squared tests (or suitable alternative) used for comparisons where applicable. Tolerability will also be evaluated, summarizing rates of dose delays or modifications, reasons patients end treatment, and time to end of active treatment.
Duration of response (DoR) | up to 2 years
  Defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a complete response or partial response to the earliest date progression is documented, or death if no prior evidence of disease progression. The distribution of DoR will be estimated using the method of Kaplan-Meier.
Overall survival (OS) | up to 2 years
  Defined as the time from randomization to death due to any cause. Patients who are alive will be censored at last follow-up for OS. The distribution of survival time will be estimated using the method of Kaplan-Meier. OS will be compared between treatment arms using the log-rank test. OS medians, survival rates and hazard ratio will be estimated along with 95% confidence intervals.
Progression free rate at 8 weeks (PFR8) | At 8 weeks
  Defined as the proportion of evaluable patients who are alive and without evidence of disease progression 8 weeks after initiation of study therapy. The final PFR8 point estimate and corresponding 95% confidence interval calculated using Clopper-Pearson method.

OTHER OUTCOMES:
CDK4 copy number | Up to 2 years
  Explore data on CDK4 copy number (by fluorescence in situ hybridization [FISH] or other molecular testing) through plots and summary statistics.
Infiltrating immune cell subsets and tumor and immune cell major histocompatibility complex (MHC) and PD-L1 expression | Up to 2 years
  Conduct multiplex immunohistochemistry using archival tumor tissue (where available) to summarize densities of infiltrating immune cell subsets and tumor and immune cell MHC and PD-L1 expression.
Relationship between CDK4 copy number and the tumor immune microenvironment and clinical outcomes | up to 2 years
  Explore the relationship between CDK4 copy number and (a) the tumor immune microenvironment as defined by multiplex immunohistochemistry and (b) clinical outcomes from study treatment Clinical endpoints include PFS, objective response rate, OS, PFR8, and DoR. Cox regression will be used on time-to-event outcomes and T-test on binary outcomes
Efficacy and toxicity endpoints | Up to 2 years
  Explore the efficacy and toxicity endpoints for patients who progress on palbociclib monotherapy and crossover to the palbociclib plus cemiplimab combination A sensitivity analysis will be conducted to see how crossover effects overall survival. Rate and severity of adverse events will be used to assess differences between crossover and non-crossover patients.

CONTACTS AND LOCATIONS:
Locations (194):
- United States (194):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Mercy Cancer Center, Merced, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin